CLINICAL TRIAL: NCT06247865
Title: Characterising Biomarkers and Clinical Algorithms to Identify Oncology Patients on Immune Checkpoint Inhibitors (ICPI) That Are at Greater Risk of Developing Immune-related Adverse Events (irAE)
Brief Title: BIO-CHECKPOINT 0 Biomarkers to Identify Oncology Patients on ICPI at Greater Risk of irAE
Status: Completed | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: PHU/2023/28
Record Dates: First submitted 2024-01-17; First posted 2024-02-08 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will collect leftover clinic blood samples on new oncology ICPI patients and test them for routine blood tests and malondialdehyde. Malondialdehyde can assess the body's oxidative stress level, a condition where your body lacks antioxidants. The NHS does not offer a malondialdehyde test presently, the study would produce a new NHS blood test. Once testing is completed the samples will be destroyed. Blood test results will be correlated to the patient's outcome i.e., did they have an irAE and assess if there are any differences in the results. From this information, the investigators hope to understand which blood tests help to highlight if a patient is at risk of developing irAE before it occurs.

DETAILED DESCRIPTION:
Immune checkpoint inhibitors (ICPI) are a type of cancer treatment. Unlike traditional chemotherapy and radiation, which damages both the cancer and the healthy tissue, ICPI targets cancer directly by altering the immune system. Cancer cells produce high levels of protein called checkpoint proteins, which bind to white blood cells (which are part of the immune system) and stops them from working. Effectively the cancer is pushing a stop button on the immune system and the body can no longer fight it off. ICPIs block and remove these cancer checkpoint proteins, which allows the immune system to target the cancer again removing this stop button.

ICPI has great success in treating cancer and 10% of oncology NHS patients receive this treatment, although this number is increasing. However, ICPI carries a risk of a type of side effect called immune related adverse events (irAE). irAEs can be life threatening and present with similar symptoms to the patient's cancer. For example, a patient may have kidney cancer and after treatment with ICPI develop kidney failure. It is difficult for the doctor to tell if this is the cancer progressing or a side effect of the treatment. Delays in diagnosing irAE can lead to unnecessary hospitalisation, unnecessary breaks in treatment, lifelong side-effects, and death.

Currently there is not a unified blood test panel for ICPI patients, and the cancer societies have produced little guidance for the doctors to use. At Portsmouth what blood tests you get as an ICPI patient depend on which clinician you see. There is also little research as researchers are focussing on using blood tests to predict ICPI treatment success rather than the chance of a patient developing an irAE.

This study intends to collect leftover blood from routine clinical blood draws from oncology patients being treated with ICPIs for the first time. The investigators will freeze the leftover samples and test them a month later for different routine blood tests as well as malondialdehyde. Malondialdehyde is a blood test that can assess the body's oxidative stress level, a condition where your body lacks antioxidants. Testing for malondialdehyde is not available in the NHS and we would produce a new NHS blood test as part of this study. Once testing is completed the samples will be destroyed as per our normal protocol. At the end of the study, blood test results will be correlated to the patient's outcome i.e., did they have an irAE or not and assess if there are any differences in their blood test results. From this information the study hopes to understand which blood tests help to highlight if a patient is at a risk of developing irAE before it occurs. It also aims to develop a new method for measuring malondialdehyde.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Oncology patients
* Who is prescribed FDA approved check point inhibitors: (ipilimumab, nivolumab, pembrolizumab, cemiplimab, atezolizumab, avelumab, and durvalumab)
* All cancer subtypes are included

Exclusion Criteria:

* <18 years of age
* Those previously been treated with checkpoint inhibitors.
* Those with a previous medical history of autoimmune disease
* Those with previous medical history of endocrine diseases
* Those with a pre-existing malignancy
* Non-Queen Alexandra hospital oncology patients
* Lacking capacity to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Oncology patients, whom have been prescribed ICPIs for the first time, will be identified via the chemotherapy scheduling system.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Prediction of patient risk of irAE. | 2 years
  A calculation or clinical flow chart that can accurately predict patient's at risk of onset of irAE using routine blood tests and novel biomarkers. Sensitivity, specificity will be calculated and ROC curves.

SECONDARY OUTCOMES:
Significant difference in any established biochemistry, haematology and immunology blood tests in those who develop irAE when compared to those that don't. | 2 years
  Significant difference (p<0.05) in blood test results (concentrations) of those who develop an irAE, opposed to those who don't. Tests include but not limited too: interleukin 6, haptoglobin, C-reactive protein, Beta 2 macroglobin, complement proteins (C3 and C3), lactate dehydrogenase, ferritin, etc.
Valid liquid chromatograph method fit for clinical laboratory use. | 2 years
  A working liquid chromatograph method fit for use in a clinical laboratory will be developed with working calibration curve and IQC's. With a defined lower limit of blank, lower limit of detection, lower limit of quantification, inter/intra-precision, etc. Calibration curve will aim to have a linearity of R=0.90.
Significance of Malondialdehyde results. | 2 years
  Malondialdehyde results will be significantly different (p<0.05) in those who develop an irAE opposed to those who do not.

CONTACTS AND LOCATIONS:
Locations (1):
- Portsmouth Hospitals NHS Trust, Queen Alexandra Hospital, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-02): https://cdn.clinicaltrials.gov/large-docs/65/NCT06247865/Prot_SAP_000.pdf